CLINICAL TRIAL: NCT05051735
Title: PARASTOP - Paracetamol With Strong Opioids. A Randomized, Double-blind, Parallel-group Non-inferiority Phase III Withdrawal Trial of Paracetamol Versus Placebo in Conjunction With Opioids for Moderate to Severe Cancer-related Pain
Brief Title: PARASTOP - Paracetamol With Strong Opioids
Acronym: PARASTOP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Ørnulf Paulsen, Senior Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180946
Record Dates: First submitted 2021-09-11; First posted 2021-09-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cancer Pain; Cancer
Keywords: Cancer Pain; Pain; Analgesics; Sensory System Agents; Physiological Effects of Drugs
MeSH Terms: conditions — Cancer Pain; Neoplasms; Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracetamol (Experimental): Paracetamol P.O. 500 mg 2 tablets four times a day for 7 days
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): Placebo P.O. 2 tablets four times a day for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — Paracetamol 500 mg
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Current guidelines recommend all people with cancer-related pain should be prescribed paracetamol, even those receiving high doses of strong pain killers (opioids) such as morphine. Although this has been shown in studies to be beneficial in other conditions, for instance dental work and after surgery, it has not been shown to further improve pain in people with cancer-related pain. Taking tablets is burdensome to patients and the study aims to determine whether the inconvenience of taking eight extra paracetamol tablets per day can be justified.

The study plans to show whether or not pain control is changed (non-inferior) when stopping paracetamol compared to continued use of paracetamol in people already taking strong pain killers for cancer-related pain. Voluntary participants who are taking a combination of paracetamol and a strong opioid are recruited to the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years of age inclusive, at the time of signing the informed consent.
* ≥50 kg (due to paracetamol dosage)
* Participants who are under palliative care or oncology service review
* Diagnosis of metastatic cancer
* Clinician-predicted life expectancy >2 months
* Receiving daily regular strong opioids for cancer pain
* Receiving stable scheduled opioid dose last 48 hours*
* Receiving paracetamol 1 gram x three or four times a day for at least five days
* Average pain intensity past 24 hours ≥ 2 and ≤ 7 (NRS 0-10)*
* Able to take study drug/placebo as tablets
* Able to comply with all study procedures
* Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

  * It is allowed to repeat procedure within the screening period without considering the participant being a rescreen

Exclusion Criteria:

* History of allergy or hypersensitivity to any of the active substances or excipients in the study drug
* Known severe liver or renal failure equivalent with CTCAE Grade 3 or 4* precluding continuation of paracetamol. (*Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0)
* Participants receiving subcutaneous, intravenous, intrathecal, or epidural opioid therapy
* Participants receiving systemic anticancer treatment during the intervention period if they are anticipated to have increasing pain or other symptoms related to the treatment
* Co-enrolment in other drug trials. Participants will not be enrolled in any other on-going interventional clinical trial. Study participants may be enrolled in non-interventional research (e.g. questionnaire, tissue collection studies)
* Previously enrolled in this study
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
To establish whether placebo with strong opioids compared to paracetamol together with strong opioids provides non-inferior analgesia for cancer-related pain. | 7 days
  Numeric Rating Scale 0-10: Average pain intensity past 24 hours

SECONDARY OUTCOMES:
To establish whether placebo with strong opioids compared to paracetamol with strong opioids changes opioid related side effects. | 7 days
  Opioid Side Effects Questionnaire
To establish whether placebo with strong opioids compared to paracetamol with strong opioids changes global rating of improvement. | 7 days
  Patient Global Impression of Change
To establish whether placebo with strong opioids compared to paracetamol with strong opioids changes opioid requirements. | 7 days
  Opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Ørnulf Paulsen, Principal Investigator — Telemark Hospital Trust
Locations (15):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
- Norway (12):
  - Vestre Viken Hospital Trust, Drammen, Drammen
  - Førde Hospital Trust, Førde, Førde
  - Østfold Hospital Trust, Sarpsborg, Grålum
  - Sørlandet Hospital Trust, Kristiansand, Kristiansand
  - Stavanger University Hospital, Stavanger, Stavanger
  - Helse Møre og Romsdal, Ålesund
  - Akershus University Hospital, Lørenskog
  - OsloUH, Oslo
  - Telemark Hospital Trust, Skien
  - Universitetssykehuset Nord-Norge, Tromsø
  - St. Olavs Hospital, Trondheim
  - Vestfold Hospital trust, Tønsberg
- Makere University Hospital, Kampala, Uganda
- Edinburgh Cancer Research, Edinburgh, United Kingdom